CLINICAL TRIAL: NCT01696188
Title: Comparison of In-Plane vs. Out-of-Plane Ultrasound-Guided Approach for Interscalene Nerve Catheters: a Prospective, Randomized Trial
Brief Title: A Study Comparing Two Methods of Placing an Interscalene Nerve Catheter for Postoperative Pain Control in Patients Who Undergo Open Shoulder Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 12D.328
Record Dates: First submitted 2012-09-13; First posted 2012-09-28 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-10

CONDITIONS: Shoulder Pain
Keywords: Interscalene; nerve block; nerve catheter; in-plane; out-of-plane; anterolateral approach; posterior approach; shoulder surgery
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- In-plane group (Experimental): This group will receive an interscalene catheter placed with in-plane approach.
  Interventions: Device: interscalene nerve catheter
- Out-of-plane group (Experimental): This group will receive an interscalene catheter with an out-of-plan approach.
  Interventions: Device: interscalene nerve catheter

INTERVENTIONS:
Device: interscalene nerve catheter
  Other Names: Peripheral nerve catheter kit, B Braun (Bethlehem, PA)

SUMMARY:
This is a randomized, double-blinded, prospective study designed to compare two approaches (in the plane of the ultrasound beam and out of the plane of the ultrasound beam) to placing an interscalene nerve block and catheter for pain control after open shoulder surgery. Both approaches have been used successfully but neither has been proven to be superior. Our endpoints are pain scores, time for block placement, and catheter dislodgements. We hypothesized that patients with the out-of-plane approach would have decreased pain and fewer catheter dislodgements.

DETAILED DESCRIPTION:
Interscalene nerve block is an effective method of analgesia for surgery of the upper extremity. Perineural interscalene catheters offer the advantage of extended pain relief up to 48 hours after shoulder surgery. This is a prospective, randomized trial designed to compare two approaches (posterior and anterolateral) to interscalene continuous nerve catheter placement for analgesia after open shoulder surgery (open rotator cuff repair, total shoulder arthroplasty or revision, hemi-arthroplasty, or proximal humerus open reduction internal fixation). Specifically, the objectives of this study are to compare measured pain scores, opioid consumption, and catheter dislodgements. We hypothesize that the anterolateral approach will produce lower pain scores, less opioid consumption, and fewer catheter dislodgements.

All patients undergoing open shoulder surgery will be recruited and enrollment in the study will not deviate from the current standard of care at Thomas Jefferson University Hospital. All nerve blocks will be placed by a regional anesthesiologist or a fellow in regional anesthesia. Patient medical history will be obtained and blocks will be placed per usual protocol. Block efficacy will be assessed by physical exam immediately after placement by the anesthesiologist and another member of the research team. Operative details, including medications given, will be recorded.

Patient pain scores and medications given in the PACU will be recorded. Supplementary analgesics will be available. Pain scores, medications given, and sensory examinations will be recorded for 48 hours postoperatively. Data will be analyzed both at the conclusion of the study and at several interims before that.

ELIGIBILITY:
Inclusion Criteria:

* speaks English

Exclusion Criteria:

* children,
* neuropathy in operative arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Fredrickson MJ, Ball CM, Dalgleish AJ. Posterior versus anterolateral approach interscalene catheter placement: a prospective randomized trial. Reg Anesth Pain Med. 2011 Mar-Apr;36(2):125-33. doi: 10.1097/aap.0b013e31820d5ee6. PMID 21425511
- [Background] Antonakakis JG, Sites BD, Shiffrin J. Ultrasound-guided posterior approach for the placement of a continuous interscalene catheter. Reg Anesth Pain Med. 2009 Jan-Feb;34(1):64-8. doi: 10.1016/AAP.0b013e3181933a53. PMID 19258990
- [Background] Mariano ER, Loland VJ, Ilfeld BM. Interscalene perineural catheter placement using an ultrasound-guided posterior approach. Reg Anesth Pain Med. 2009 Jan-Feb;34(1):60-3. doi: 10.1097/AAP.0b013e3181933af7. PMID 19258989

RESULTS

PARTICIPANT FLOW:
Groups:
- In-plane Group: This group will receive an interscalene catheter placed with in-plane approach.
  interscalene nerve catheter
- Out-of-plane Group: This group will receive an interscalene catheter with an out-of-plane approach.
  interscalene nerve catheter
Period: Overall Study
Arm/Group | In-plane Group | Out-of-plane Group
Started | 41 | 43
Completed | 40 | 42
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Out-of-plane Group: This group will receive an interscalene catheter with an out-of-plan approach.
  interscalene nerve catheter
- Total: Total of all reporting groups
Arm/Group | In-plane Group | Out-of-plane Group | Total
Number analyzed (Participants) | 40 | 42 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (10.7) | 63.8 (12) | 65.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 17 | 42
  Male | 15 | 25 | 40
Region of Enrollment [Number; unit: participants]
  United States | 40 | 42 | 82

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale Pain Scores
Description: Pain was rated from 0 (no pain) to 10 (worst pain imaginable)
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | In-plane Group | Out-of-plane Group
Number analyzed (Participants) | 40 | 42
units on a scale | 1.3 [0 to 3.8] | 1.5 [0 to 4.5]

2. Secondary Outcome: Catheter Dislodgements
Description: Inspect the peripheral nerve catheters at 24 hours postoperatively and assess for being in-place or not.
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | In-plane Group | Out-of-plane Group
Number analyzed (Participants) | 40 | 42
participants | 4 | 1

3. Secondary Outcome: Opioid Consumption
Description: Calculate the total amount of opioid consumed in the first 48 hours after surgery using a standard opioid conversion scale. 1 mg hydrocodone = 0.33 mg IV morphine, 1 mg oxycodone = 0.50 mg morphine IV, 1 mg hydromorphone PO = 1.33 mg morphine IV, 1 mcg fentanyl = 0.1 mg morphine IV, 1 mg hydromorphone IV = 6.67 mg morphine IV
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: mg IV morphine equivalents
Arm/Group | In-plane Group | Out-of-plane Group
Number analyzed (Participants) | 40 | 42
mg IV morphine equivalents | 25.0 [12.5 to 65.0] | 35.3 [24.8 to 70.7]

4. Secondary Outcome: Time for Block Placement
Description: Calculate the time to perform the nerve block procedure.
Time Frame: immediately post-procedure
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | In-plane Group | Out-of-plane Group
Number analyzed (Participants) | 40 | 42
seconds | 296 [255 to 337] | 257 [238 to 277]

ADVERSE EVENTS:
Arm/Group | In-plane Group | Out-of-plane Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42
Other Adverse Events (participants affected / at risk) | 0/40 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes